CLINICAL TRIAL: NCT00712972
Title: Evaluation of the Effectiveness of the Medial Parapatellar Knee Injection Technique
Brief Title: Evaluation of the Medial Parapatellar Knee Injection Technique
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Harold L Battenfield / Dr., Oklahoma State University
Other Study IDs: IRB#200808
Record Dates: First submitted 2008-07-08; First posted 2008-07-11 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis; Accuracy of Intraarticular Needle Placement
Keywords: knee injection; parapatellar
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients enrolled in this study are those whom present to our institution for elective knee arthroscopy. All patients scheduled to receive a knee arthroscopy scheduled through the office of Dr. Harold Battenfield will be asked to participate in the study on the day of their procedure as long as they do not fall into one of the exclusion criteria categories.
  Patients will not be allowed to participate in this study if they have an allergy to iodine or shell fish, if they have a knee effusion diagnosed clinically on the day of surgery, if the knee or surrounding tissues display cellulitis or other signs of infection, or if the patient has had a traumatic accident to their knee which significantly changes its anatomical relationships

SUMMARY:
The goal of our study is to present important anatomic considerations which should be considered before knee injection is performed. Additionally, we have developed important procedural augments to the traditional para-patellar injection techniques in order to exceed the accuracy and safety previously reported for the infra-patellar approaches We have developed an injection technique which mechanically is similar to current techniques practiced and poses no additional risks or discomfort to the patient. The basis of our technique and its success is through recognition of anatomic factors and avoidance of possible iatrogenic injuries which exist when using other knee injection technique. The focus of our study is to validate the clinical accuracy we have been obtaining using our technique through fluoroscopically confirmed visualized confirmation of repeated intra-articular deposit. Additionally we want to document the range of needle length we require to properly access the knee joint in our population to substantiate the importance of needle length. Needle length is a critical factor in obese patients whom have larger infra-patellar fat pads.

Our hypothesis is that when using a 6 inch 22 gage needle for intra-articular knee injections through the medial joint line approach, while utilizing the medial wall of the lateral femoral condyle as an intra-articular stop point for needle insertion, the accuracy of intra-articular deposit will exceed the values currently reported in the literature which is approximately 75% success rate.

To prove this point we will be injecting 2 cc of radiocontrast dye into the joint space and than immediatly view the joint flouroscopicly after the knee has been brought through 10 cycles of flexion and extension.

DETAILED DESCRIPTION:
Injection into the knee joint, although considered a remedial procedure by much of the medical community, is not as easy a procedure to reproducibly and accurately perform as one would believe. Numerous authors have estimated that between 20 to over 30 percent of knee injection procedures fail to deposit the injectate into the joint space (6),(7),(9) (11). In response to the reportedly high complication rates associated with intra-articular deposit of injectate, numerous authors have published different techniques, injection sites, and tricks to help the clinician. Techniques such as air arthrography (12)(13), the backflow technique (7), the triangle technique (11), and others have added complexity and time to a seemingly easy procedure.

Specific anatomic relationships within the knee joint provide larger access windows and relatively easier entry for some techniques than for others. Additionally, the presence of hyaline articular cartilage, the smooth, nonreplicable joint surface integral to the efficient and pain free articulation of joints adds another complexity and concern in access to the knee joint. Iatrogenic damage to this cartilage is probable with some commonly employed injection techniques. Damage to the articular surface is the anatomic equivalent of arthritic pathologic change within the knee joint.

Much of the confusion surrounding accurate intra-articular injection stems from the anatomic relationships we are taught during our training. Anatomical atlases depict the layers of the knee joint in such a fashion as there being a tangible and recognizable joint space to easily insert a needle. This is not the case in the normal knee which does not have a knee effusion. The reality is that the normal adult knee has 2 cc of synovial fluid dispersed as an extremely thin film over the top of the articular cartilage. The synovial membrane in effect rests directly on top of the articular cartilage and hence the joint space is actually a potential space. Even though this is the case, there are three predominate areas of recess within the knee joint where if the needle is accurately placed, this potential space can be developed. These three regions are the inter-trochlear groove, inter-condylar notch, and the suprapatellar pouch.

The inter-trochlear groove is the region on the anterior surface of the femur which lies directly below the patella when the knee is in its extended position. The inter-trochlear groove is covered with articular cartilage which is integral in maintaining normal pain free patellofemoral articulation.

The inter-condylar notch is a region of the femur on its most distal aspect which houses the ACL and PCL tendons. The inter-condylar notch is not an articular region of the knee joint and is not covered with articular cartilage. The fact that there is no articular cartilage in the inter-condylar notch significantly reduces chances of iatrogenic cartilage damage. Placement of the needle precisely into one of these spaces is crucial for a successful injection.

There has been debate as to the safest and most reliable technique for intra-articular knee injections over the last decade. Five common procedures, including the technique studied in this research protocol are currently employed by the medical community for access into the knee joint. These five techniques all share the same basic materials and principles, and all five carry the same risks associated with insertion of a foreign body into a joint space.

The medial and lateral infra-patellar techniques are the first two techniques considered. Regardless of the side of the knee the needle is placed into, the infra-patellar technique positions the needle between the patella and the femur while the knee is in the extended position on the examination table. The infra-patellar injection technique uses a needle endpoint position which lies within the intertrochlear groove.

The medial and lateral joint line techniques, also known as the para-patellar techniques are other commonly utilized techniques. The para-patellar injection techniques route of entry into the knee joint is through the soft spot just proximal to the tibial plateau, on either the medial or lateral side of the patellar ligament. In the para-patellar injection techniques needle insertion is performed while the knee is flexed to 90 degrees off the edge of the examination table and the end point is within the intercondylar notch.

The last injection site occasionally used, orientates the needle into the suprapatellar pouch. This route of injection is at times chosen due to the fact that it is a reliable region to aspirate a knee when there is a large effusion. Although the suprapatellar pouch is the largest potential space in the knee joint, this space is essentially closed down in the knee which lacks an effusion. Successful injection into the suprapatellar pouch is analogous to perfect placement of a needle between two sequential pages in a book. When no joint effusion is present, this space lacks any tactile stimulus to indicate proper needle orientation and depth, and hence successful injections from this route are difficult and unreliable.

Another issue plaguing current knee injection practices is the choice of needle used. The vast majority of medical offices stock 1.5 inch long needles as this is by far the most common production length available. Obviously other lengths are available, yet they are more of a special order type item which is not on hand at the time of the knee injection. Needle length is not a consideration to nearly all practitioners whom are performing knee injections. This is partially due to the anatomic misconceptions of the intra-articular space as a wide open and easily accessible region as depicted in anatomy texts. When injecting into a knee using the para-patellar technique there are important structures the needle must pass through before it will enter into the synovial space. Structures such as pre-patellar bursal tissue, subcutaneous adipose, fascia, the infrapatellar fat pad, and possibly hypertrophic thickened synovium are distinct anatomic structures which vary in depth and can quickly use up the working length of a standard needle before it is able to access the intra-articular space. With the growing obesity problem in America, the issue of adequate needle length is becoming an increasingly important consideration.

The current literature regarding knee injections does not seem to account for required needle length. Numerous studies, including the ones referred to in this protocol utilize needles which are 2 inches in length or less, and these same studies report a low accuracy of intra-articular penetrance with techniques which transverse the infra-patellar fat pad (1),(2),(6).

The need for accurate placement of a substrate directly into the knee joint has increased over the last few years as the popularity of proteoglycan hyaluronic acid (HA) preparations are growing in popularity for treatment of osteoarthritis (OA). Unlike steroid injections largely utilized in the past for symptomatic treatment of OA, the HA preparations for efficiency require accurate placement within the synovial pocket of the knee joint. Briefly this difference is based upon the mechanism of action of these two macromolecules. Steroids function as anti-inflammatory mediators, inhibiting the ability for recruitment and entry of inflammatory cells into the knee joint. Because of this, inaccurate deposit of steroid injections in a peri-articular location will still result in clinical benefits through a paracrine mechanism (7),(8). HA preparations are made of proteoglycans, which are large negatively charged protein polysaccharide molecules, which recruit water into the joint space and articular cartilage. Proteoglycans function like a sponge by providing hydrodynamic cushioning to the joint during weight bearing . Unlike steroid a preparation, if HA is mistakenly injected into the peri-articular soft tissues, its clinical benefit is essentially nullified (1), (6),(10). In relation to the above discussion on proper needle length, inadvertent placement of HA into the infra-patellar fat pad as a result of too short of a needle will result in the injected material to remain within the fat pad, unable to reach the intra-articuar space where it will be effective. In a 5 subject MRI evaluation of the size of the infra-patellar fat pad, Jackson et al. has shown size variations ranging from 1.8 to 2.2 inches between the skin and articular surface (1). Obviously a larger sample size is required to achieve a more accurate distribution of pre-articular soft tissue mass but this reported range does add validity to the importance of needle size.

Current hyaluronic acid preparations involve a series of 3-5 injections and currently have a clinical effectiveness for pain relief for approximately 50% of patients receiving the series of injections. Although this study is not intended to test or evaluate the above clinical efficacy of HA, the fact that the HA injectate may be mistakenly deposited into the infrapatellar fat pad secondary to improper needle length or poor technique may be an important factor in its low clinical effectiveness.

Recently authors such as Jackson (1), Wind (2) Toda (6), and others have reported excellent success with intra-articular injections through the infra-patellar approach to the knee. Their studies have touted the high accuracy in delivering a substrate into the intra-articular space. Additionally their work has shown considerably lower accuracy in intra-articular deposit via one of the joint line approaches. Their articles have set a precedent in the medical community for the infra-patellar injection approach.

The biggest concern we have with the infra-patellar approach is centered on damage to the articular cartilage of the inferior surface of the patella as well as the trochlear groove of the femur. There is very limited space between the patella and the femur in the joint which lacks an effusion. MRI evaluation of a normal knee joint displays at most 1 - 2 mm of potential space where a needle can be inserted into to provide a joint injection without damage to articular cartilage. Radiographs provide a false interpretation of available free space at the patellofemoral joint. Indeed the articular cartilage which resides in this joint is very thick producing the radiolucent clear region appreciated on radiographs. The normal thickness of articular cartilage on the condyles is 4.0 and 3.7 mm for the medial and lateral sides respectively. The normal thickness of articular cartilage on the patella is 5 mm in depth and holds the distinction of being the thickest layer of articular cartilage in the body (3). The correct placement of the injection needle is further complicated by two additional factors, one being no specific palpable entry point to insert the needle into. A lack of a definitive palpable entry point results in estimation and clinical experience to provide the initial starting point. Secondly, with the infra-patellar injection site there is no definitive palpable end point to aid in stopping the insertion of the needle. This lack of end point unfortunately results in excessive insertion of the needle with iatrogenic articular trauma produced by the cutting edge of the needle tip.

A second consideration associated with the reported successful nature of intra-articular dissemination through the infrapatellar approach concerns the "blowout" force generated by hydrodynamic pressures. Because no definitive end point of needle insertion in this region exists until after the needle tip has traversed the articular cartilage surface, forceful injection, even with some pre-emptive needle withdrawal, will cause the dye to initially be forced into the articular cartilage substrate before it can be extravisated out into the articular space. This forced evacuation out through the cartilage is due to the molecular structure of hyaline cartilage, its collagen fiber orientation, and its resultant resilience to surface shear forces. Indeed the collagen fiber network restricts absorption of fluid to only 20% of the cartilage's potential volume, all other fluid will resultantly be forcefully evacuated from the extra cellular matrix into the joint space. (4) a fluid bolus of a couple of cc results in the cartilage's inability to retain the fluid in its extracellular matrix resulting in a "blowout" of the artiticular surface to allow release of the material into the joint space. Although this forceful extravisation provides fluoroscopic evidence of successful fluid bolus placement into the joint space, it does so at the cost of the integrity of the articular cartilage at the injection site. This is in contrast to the accommodating, compliant, and hydrophobic nature of adipose tissue in the infrapatellar fat pad which tends to expand around an injected fluid bolis and retain the injected substrate resulting in failed intra-articular deposit.

The above observations suggest that although the infra-patellar approach does effectively provide for a means of injection into the knee joint's space, it does so at a cost to the articular cartilage which in this author's opinion is an unnecessary risk and complication. When one considers that the common HA preparations on the market today require between 3 - 5 total injections, and the fact that repeat intra-articular treatments are often provided on a biannual basis, the potential for iatrogenic injury quickly multiplies.

The goal of our study is to present important anatomic considerations which should be considered before knee injection is performed. Additionally, we have developed important procedural augments to the traditional para-patellar injection techniques in order to exceed the accuracy and safety previously reported for the infra-patellar approaches.

This study is not intended to directly compare our results against those achieved in the infra-patellar technique, this research does not refute the excellent clinical results achievable through the infra-patellar techniques. The intention of this study is to show that utilizing our specific technique for para-patellar knee injection we can achieve accurate intra-articular deposit over 95% of the time, which is a considerable improvement over previously reported results using the para-patellar approach (1). Additionally our technique avoids the theoretical iatrogenic injury associated with the infra-patellar approach.

We have developed an injection technique which mechanically is similar to current techniques practiced and poses no additional risks or discomfort to the patient. The basis of our technique and its success is through recognition of the factors mentioned above. The focus of our study is to validate the clinical accuracy we have been obtaining using this technique through fluoroscopically confirmed visualized confirmation of repeated intra-articular deposit. Additionally we want to document the range of needle length we require to properly access the knee joint in our population to substantiate the importance of needle length. Needle length is a critical factor in obese patients whom have larger infra-patellar fat pads All intra-articular injection will be performed by, Drs Harold Battenfield and Brian Drake. The study population will be equally divided between the two such that each investigator will inject an even number of knees. The distribution of the patients to each physician will be randomized based upon time of presence. Drs Battenfield and Drake will alternate "turns" where the first patient will be injected by one physician than the next sequential patient will be injected by the other physician until a significant number of injections have been performed The study population will consist of patients already receiving a knee arthroscopy at our institution. It is important to note that the study information will be kept completely separate and isolated from the operative patient chart. All involved patients will be issued a study number and any information recorded will be done so under that number. All patients involved in the study will have their sex, height, weight, and success of attempted insertion recorded. No names, no birthdates, no medical record numbers, nor any other specific and identifiable information will be recorded.

This entire procedure will be performed after the patient has been administered the general anesthesia as is customary during a knee arthroscopy. The injection protocol adds less than 2 minutes to the surgical time of the arthroscopy.

In order to test our hypothesis we will draw up 2 cc of radiopaque dye (Isovue dye) into a 5 cc syringe attached to a 6 inch 22 gage spinal needle utilizing sterile technique. This injection is performed on the same knee as is scheduled for arthroscopy. The patient will be positioned into the standard arthroscopy leg immobilizer which allows the leg to hang dependently in a 90 degree flexed position, which mimics the typical position as would be experienced in the office.

The anatomic location for needle penetration is easily found in even obese patients by simple digital palpation of the "soft spot" which exists directly above the tibial plateau. This soft spot will then be marked with a small blunt object. We will use a "clickable" retractable ink pen while the ink cartage is in its retracted position to provide a nice "bullseye" demarcation on the skin surface.

Once the site is marked the skin surface will be cleansed with a betadine based prepping solution utilizing sterile technique.

The needle will be inserted through the predemarcated site, and the trajectory of the needle will be directed toward the medial wall of the lateral femoral condyle, within the inter-condylar notch. Insertion of the needle will proceed until confirmed tactile impact against the condyle is achieved. The depth the needle inserted into the skin will then be sterilely marked on the needles shaft with a sterile marking pen, and this length is later measured. Without retraction of the needle the 2 cc of radiopaque dye will then be injected into the knee joint.

The injection volume of 2 cc is chosen based upon the fact that this is the volume of fluid commonly packaged into viscosupplimentation (hyaluronic acid) preparations. The 2cc volume will more closely correlate with in office injection conditions.

Once the dye is successfully placed within the joint, and the needle removed, the joint will than be flexed and extended a total of 10 revolutions ending in an extended position. This flexion and extension cycling provides an opportunity for intra-articular injectate to disseminate around the joint's surface.

At this point mobile fluoroscopy will be utilized to visualize the knee in both the AP and Lateral planes. Evaluation of proper placement of the dye is confirmed by noting the extravasation characteristics of the dye fluoroscopically. Successful injection into the joint space is anticipated to result in uniform distribution of the dye along the margins of the femoral condyles, evenly coating the joint surface as previously reported by Jackson (1), Wind(2), and Toda(6).

In contrast, if radiopaque dye is injected into the fat pad an entirely different radiographic image will result. The infra-patellar fat pad acts as an anatomic "cork" preventing materials injected into its substance from entering into the knee joint where it is intended to go. If the needle does not penetrate the synovial membrane than there is a low likelihood of extra-articular material from entering the knee joint. This is a normal anatomic phenomena that our bodies utilize to help prevent intra-articular infections. The joint space is in effect a protected region of the body, much like the central nervous system is protected by the blood brain barrier. If our injection technique inaccurately places the radiopaque dye into the infra-patellar fat pad, the result will be a well circumscribed radiopaque "blob" which sits extra-articularly and is easily recognized by the post-injection floroscopy. Authors such as Jackson (1), Wind (2), and Toda (6) have shown the accumulation phenomenon of injected substrate into the infra-patellar fat pad With this procedure complete, the patient's leg will be prepped and draped in the normal standard manner and the arthroscopy will be carried out as would normally be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in this study are those whom present to our institution for elective knee arthroscopy. All patients scheduled to receive a knee arthroscopy scheduled through the office of Dr. Harold Battenfield will be asked to participate in the study on the day of their procedure as long as they do not fall into one of the exclusion criteria categories

Exclusion Criteria:

* Patients will not be allowed to participate in this study if they have an allergy to iodine or shell fish, if they have a knee effusion diagnosed clinically on the day of surgery, if the knee or surrounding tissues display cellulitis or other signs of infection, or if the patient has had a traumatic accident to their knee which significantly changes its anatomical relationships

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in this study are those whom present to our institution for elective knee arthroscopy. All patients scheduled to receive a knee arthroscopy scheduled through the office of Dr. Harold Battenfield will be asked to participate in the study on the day of their procedure as long as they do not fall into one of the exclusion criteria categories.
  The patient population often encountered in our practice includes a variety of patient demographics. We enjoy patient referrals from numerous primary care physicians in the community as well as through Oklahoma State University Medical Center's emergency department. Additionally we work closely with one of the regions primary workers compensation agencies. Because of our numerous referral resources, our patient population is considerably varied and provides an ample mixture of patient demographics to allow us to reasonably extrapolate and compare our study results to the general population
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The percentage of successfull intra-articular deposits of radiocontrast dye into the knee joint using our medial parapatellar joint line approach and comparison of this value to previously reported values in the literature | one year

SECONDARY OUTCOMES:
The length of the needle which is required to successfully transverse the infrapatellar fat pad in order to deposit injectate into the knee joint | one year

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Battenfield, D.O., Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University Collage of Health Sciences, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Jackson DW, Evans NA, Thomas BM. Accuracy of needle placement into the intra-articular space of the knee. J Bone Joint Surg Am. 2002 Sep;84(9):1522-7. doi: 10.2106/00004623-200209000-00003. PMID 12208907
- [Background] Wind WM Jr, Smolinski RJ. Reliability of common knee injection sites with low-volume injections. J Arthroplasty. 2004 Oct;19(7):858-61. doi: 10.1016/j.arth.2004.02.042. PMID 15483801
- [Background] Toda Y, Tsukimura N. A comparison of intra-articular hyaluronan injection accuracy rates between three approaches based on radiographic severity of knee osteoarthritis. Osteoarthritis Cartilage. 2008 Sep;16(9):980-5. doi: 10.1016/j.joca.2008.01.003. Epub 2008 Mar 12. PMID 18339561